#### Clinical Study Protocol Drug Substance NA Study Code D1843R00254 Edition Number 2

Date

October 17, 2016

# in Diabetes Mellitus (ENGAGE-DM): ENhancing outcomes through Goal Assessment and Generating Engagement

with diabetes negotiated interviewing on disease control and medication adherence in patients A 12-month study of the impact of combined shared-decision making and brief

| The second state of the second | Administrative Date of Administrative Local Administrative Date of Local Administrative Change No. Change No. | Sponsor: The following Amendment(s) and Administrative Changes have been made to this protocol since the date of preparation: Amendment No. Date of Amendment Local Amendment No: Date of Local Amendment |
|---|---|---|
| | Date of Local Administrative Change | is protocol since the date of Date of Local Amendment |

without providing advance notice to AstraZeneca and opportunity to object. This submission document contains confidential commercial information, disclosure of which is pronibited

compliance with prevailing laws and regulations. disclosed and/or published according to the AstraZeneca Global Policy on Bioethics and in Standard procedures. The clinical study protocol is publicly registered and the results are This Clinical Study Protocol has been subject to a peer review according to AstraZeneca

#### PROTOCOL SYNOPSIS

on disease control and medication adherence in patients with diabetes impact of combined shared-decision making and brief negotiated interviewing Engagement in Diabetes Mellitus (ENGAGE-DM): A 12-month study of the ENhancing outcomes through Goal Assessment and Generating

| _ |
|---------------|
| - 3 |
| rin |
| _ |
| C |
| _ |
| ă |
| 20 |
| - |
| _ |
| E |
| _ |
| ~ |
| esti |
| 9 |
| - |
| ᆵ. |
| Ø |
| 200 |
| = |
| $\overline{}$ |
| 2 |
| ~ |
| • • |

# Study site(s) and number of subjects planned

study. The Privacy Board of Horizon Blue Cross Blue Shield of New Jersey has approved this that collaborate with Horizon BCBSNJ. There are no investigational drugs being used in this number of Patient-Centered Medical Homes (PCMHs) and other population health programs New Jersey (BCBSNJ). We plan to primarily include participants who receive care in a study protocol. This prospective study will include 1,400 beneficiaries of Horizon Blue Cross Blue Shield of

| Study period | | Phase of development |
|------------------------------------------|---------|----------------------|
| Estimated date of first subject enrolled | Q3 2016 | N/A |
| Estimated date of last subject completed | Q2 2017 | N/A |

#### Study design

adherence barriers, and the benefits of maintaining blood glucose control. treatment options, goals, and preferences, medication adherence, strategies for reducing consent to engage in at least 4 telephonic discussions with pharmacists about their diabetes pharmacists. After receiving the decision aid, these patients will be asked to provide informed intervention will be mailed a patient decision aid to help prime them for encounters with medication adherence compared with usual care. Briefly, all patients allocated to the combining shared-decision making and brief negotiated interviewing on disease control and disease, we will examine the effect of pharmacist-delivered patient engagement techniques In this study of patients on at least one oral hypoglycemic therapy with poorly controlled

machine learning approaches. The use of predictive analytics will provide policy-relevant predictive analytic techniques will include logistic regression, boosted regression, and sociodemographic, clinical, medication use, and other motivational characteristics. These treatment response could be predicted based on patient characteristics, such as After the completion of the study, we will also use predictive analytics to examine whether

real-world practice. information about who is most likely to benefit from these patient engagement techniques in

#### **Objectives**

| Primary Objective: | Outcome Measures: |
|---|---|
| To examine whether a two-stage process of | Glycosylated hemoglobin (HbA1c): |
| shared decision-making and behavioral interviewing improves glycosylated | Primary outcome: Pre- to post-intervention change in mean HbA1c levels |
| nemoglobin (HbA1c) control and medication adherence among patients who have poorly- | <ul> <li>Mean levels in each study arm in the follow-<br/>up period</li> </ul> |
| COMMONIA MINOCKO. | - Proportion of patients in each study arm achieving optimal HbA1c control in the |
| | Medication adherence: |
| | <ul> <li>Continuous proportion of Days Covered<br/>(PDC) in each study arm in the follow-up</li> </ul> |
| | - Proportion of patients in each study arm |
| | the follow-up period |

| Secondary Objective: | Outcome Measure: |
|---|---|
| To develop prediction models and examine | Predictive statistics: |
| their ability to predict response to the study | <ul> <li>Cross-validated C-statistics (discriminative</li> </ul> |
| intervention based on baseline patient | ability of the model) |
| characteristics, such as sociodemographic, clinical, and medication use characteristics, as | - Cross-validated R-squares (explained |
| well as initial receptiveness to changing health | variation in treatment response) |
| behaviors. | |

| Safety Objective: | Outcome Measure: |
|-------------------|------------------|
| N/A | N/A |

#### Target subject population

age, are using at least one oral hypoglycemic agent, are not currently on insulin, and whose including non-insulin injectables. HbA1c values indicate poor disease control (≥8%). Patients may be on multiple medications, We will examine commercially-insured patients from Horizon BCBSNJ who are ≥18 years of

#### **Duration of treatment**

control group and followed for the same duration of time. diabetes control, goals and preferences. Seven-hundred patients will also be identified for a interactions with pharmacists using the two patient engagement techniques to discuss their follow-up, the patients in the intervention group will be invited to receive repeated 'booster' 700 patients will be identified for the intervention and then followed for 12 months. During

# Investigational product, dosage and mode of administration

being tested in this study. outcomes and medication adherence. There are no investigational pharmaceutical products N/A — we are examining the effect of a quality improvement intervention on diabetes

#### Statistical methods

We will use generalized estimating equations to compare the changes. programs. This laboratory information will be used to measure the change in HbA1c levels information from over 200 patient-centered medical homes and other population health levels from identification to the end of follow-up. Horizon BCBSNJ receives laboratory The primary outcome of interest will be the pre- to post-intervention change in mean HbA1c

available to them during follow-up. We will also measure and examine other adherence and the proportion of days covered (PDC), or the proportion of days that patients had medication continuous outcomes will be assessed using linear regression. medication availability. Dichotomous outcomes will compared using logistic regression, and proportion of patients achieving optimal adherence (defined by ≥80% PDC), and gaps in persistence measures as secondary outcomes, including mean PDC in each study arm, the be measured by pharmacy claims and their filling patterns. Adherence will be assessed using patients who achieved a HbA1c <8.0%. Patients' adherence to their diabetes medications will proportion of patients achieving optimal glycemic control, defined as the proportion of outcomes. The secondary glycemic outcomes will include mean HbA1c levels and the Secondary outcomes will include both glycemic outcomes and medication adherence

boosted regression and machine learning approaches. be assessed using model discrimination and performance measures, using logistic regression, the pharmacist-delivered telephonic intervention. These predictive ability of these models will medication use and adherence, other self-reported motivational characteristics, and receipt of could have been predicted based on patient factors, such as sociodemographic, clinical After study completion, we will use predictive analytics to examine whether the outcomes

#### TABLE OF CONTENTS

PAGE

| 3E |
|-----------|
| CONTENTS5 |

| | TITLE PAGE1 |
|---|---|
| | PROTOCOL SYNOPSIS2 |
| | TABLE OF CONTENTS5 |
| | LIST OF ABBREVIATIONS AND DEFINITION OF TERMS8 |
| 1. | INTRODUCTION9 |
| 1.1 | Background and rationale for conducting this study9 |
| 1.2 | Rationale for study design, doses and control groups10 |
| 1.3 | Benefit/risk and ethical assessment16 |
| 1.4 | Study Design |
| 2. | STUDY OBJECTIVES18 |
| 2.1 | Primary objective |
| 2.2 | Secondary objectives |
| 2.3 | Safety objectives |
| 2.4 | Exploratory objectives19 |
| ω | SUBJECT SELECTION, ENROLMENT, RESTRICTIONS, DISCONTINUATION AND WITHDRAWAL19 |
| 3.1 | Inclusion criteria |
| 3.2 | Exclusion criteria |
| 3.3 | Subject enrollment |
| 3.4<br>3.4.1 | Criteria for withdrawal22 Withdrawal of the informed consent22 |
| 3.5 | Discontinuation of the study22 |
| 4. | STUDY PLAN AND TIMING OF PROCEDURES23 |
| 4.1 | Enrollment/screening period23 |
| 4.2 | Treatment period |
| 4.3 | Follow-up period23 |
| 5. | STUDY ASSESSMENTS24 |
| 5.1 | Efficacy assessments24 |
| 5.2 | Safety assessments24 |
| 5.3 | Other assessments24 |

| Ethics and regulatory review39 | 10.3 |
|---|---|
| Subject data protection39 | 10.2 |
| Ethical conduct of the study39 | 10.1 |
| ETHICAL AND REGULATORY REQUIREMENTS39 | 10. |
| Data management by Brigham and Women's Hospital/Partners Healthcare and Horizon Analytics38 | 9.4 |
| Study timetable and end of study37 | 9.3 |
| Archiving of study documents | 9.2.3<br>9.2.4 |
| Monitoring of the study | 9.2<br>9.2.1<br>9.2.2 |
| Training of study site personnel36 | 9.1 |
| STUDY AND DATA MANAGEMENT36 | 9. |
| Methods for statistical analyses36 | 8.5 |
| Outcome measures for analyses36 | 8.4 |
| Definitions of analysis sets | 8.3 |
| Sample size estimate | 8.2 |
| Statistical considerations30 | 8.1 |
| STATISTICAL ANALYSES29 | .8 |
| INVESTIGATIONAL PRODUCT AND OTHER TREATMENTS29 | 7. |
| Study governance and oversight | 6.8 |
| Management of IP related toxicities | 6.7 |
| Pregnancy | 6.6 |
| Overdose | 6.5 |
| Reporting of serious adverse events26 | 6.4 |
| Recording of adverse events25 | 6.3 |
| Definitions of serious adverse event25 | 6.2 |
| Definition of adverse events | 6.1 |
| SAFETY REPORTING AND MEDICAL MANAGEMENT24 | 6. |
| Biomarker analysis | 5.6 |
| Pharmacodynamics24 | 5.5 |
| Pharmacokinetics | 5.4 |
| ical Study Protocol 3 Substance NA y Code D1843R00254 ion Number 2 October 17, 2016 | Clinical Study Protocol<br>Drug Substance NA<br>Study Code D1843R00;<br>Edition Number 2<br>Date October 17, 2016 |

| LIST OF APPENDICES | LIST OF |
|---|---|
| Schematic of analytic plan3 | Figure 3 |
| ENGAGE-DM study flowchart1 | Figure 2 |
| Schematic of the study design and patient identification | Figure 1 |
| LIST OF FIGURES | LIST OF |
| Justification: Adherence power calculation parameters and ranges3 | Table 6 |
| Justification: A1c power calculation parameters and ranges30 | Table 5 |
| Timing of study interventions2: | Table 4 |
| Patient exclusion criteria22 | Table 3 |
| List of hypoglycemic agents for inclusion2 | Table 2 |
| Patient inclusion criteria2 | Table 1 |
| LIST OF TABLES | LIST OF |
| LIST OF REFERENCES4 | 11. L |
| Audits and inspections4 | 10.6 A |
| Changes to the protocol and informed consent form3 | 10.5 C |
| Informed consent3 | 10.4 Ir |
| otocol<br>JA<br>3R00254 | Clinical Study Protocol Drug Substance NA Study Code D1843R00254 Edition Number 2 Date October 17 2016 |

Appendix A

Signatures

# LIST OF ABBREVIATIONS AND DEFINITION OF TERMS

The following abbreviations and special terms are used in this study Clinical Study Protocol.

| Abbreviation or special term | Explanation |
|------------------------------|-------------------------------------------|
| AE | Adverse event |
| GCP | Good Clinical Practice |
| ICH | International Conference on Harmonization |
| IP | Investigational Product |
| IVRS | Interactive Voice Response System |
| LSLV | Last Subject Last Visit |
| PDC | Proportion of Days Covered |
| SAE | Serious adverse event |
| T2DM | Type 2 Diabetes Mellitus |

#### 1. INTRODUCTION

# Background and rationale for conducting this study

control is common, leading to preventable complications such as stroke, heart disease, and billion in 2007, with \$58 billion spent on preventable complications. kidney failure. In the United States alone, diabetes-related health expenditures exceeded \$174 (T2DM). Although medications can effectively reduce high blood glucose levels, poor disease Both developed and developing countries face a growing epidemic of type 2 diabetes

intensify therapy, the patient's non-adherence to prescribed medications, the patient's unwillingness to accept new treatments or a combination of these factors.<sup>2,3</sup> There is growing evidence supporting several different patient-targeted interventions that could be employed in clear whether the problem is attributable to the healthcare provider's failure to appropriately additional therapy. However, among patients with poorly controlled T2DM, it is often not reductions in weight, blood pressure or glycated hemoglobin (HbA1c), and might benefit from are the mainstay of therapy for many T2DM patients, but many do not achieve the optimal changes and drug therapy. Treatment with medications such as oral antidiabetic drugs (OADs) this exceptionally common situation. T2DM is a progressive disease and treatment of T2DM comprises a combination of lifestyle

Shared decision-making (SDM) is a patient-centered approach to improve the quality of care of patients with diabetes and other chronic conditions.<sup>4</sup> SDM describes the collaborative choices more consistent with informed values; and d) greater participation in and improvement of decision making.<sup>8</sup> a) improved knowledge of options; b) more accurate expectations of benefits and harms; c) could be used to facilitate treatment choices that is in keeping with a patient's own goals.<sup>5-7</sup> A integrates both the current medical evidence and the patient's needs and preferences, and 2014 Cochrane review found that shared decision-making, supported by decision aids, led to: process where treatment decisions are made in a two-way exchange of information that

interviewing as its theoretical foundation and has shown promising results in improving adherence in other settings. <sup>13-15</sup> about how to improve their own care. For example, Brief Negotiated Interviewing (BNI), decision about treatments is made, the management of a chronic disease, such as T2DM, health risks and treatment options. 9-12 This type of interviewing technique has motivational incorporates an active listening model of counseling to facilitate patients' evaluation of their longitudinally and repeatedly, but are not necessarily designed to help patients make decisions interviewing techniques, such as motivational interviewing, are typically delivered frequently requires ongoing follow-up and patient engagement. By contrast, behavioral While shared decision-making is often employed at a single time point in time when a discrete

are complementary patient engagement techniques, no data are available on the effectiveness improve adherence to chronic disease medications. <sup>16</sup> In this spirit, even though SDM and BNI engagement, have been shown to be some of the most effective interventions available to Multi-component pharmacist-delivered interventions, particularly those rooted in patient

Date October 17, 2016 Study Code D1843R00254 Drug Substance NA Clinical Study Protocol Edition Number 2

invaluable information to healthcare providers, decision-makers and insurers to improve cost-effective (especially compared with in-person delivery), and innovative will provide techniques. Evaluating these techniques in tandem in a telephonic manner that is scalable, addition, few studies have used telephonic methods to deliver either of these behavioral of combining these 2 intervention approaches – especially in the management of T2DM. In diabetes management.

about the effectiveness of these patient engage techniques, but also about how to effectively disseminated, the results of this study will provide multiple benefits to stakeholders, not only information about which patients will benefit from the intervention moving forward. Once initial receptiveness to changing health behaviors. These findings will provide valuable characteristics, such as sociodemographic, clinical, medication adherence characteristics, and examine whether patients' response could have been predicted based on patient target patients in real-world settings. After the study is completed, the second phase of the project will use predictive analytics to

# Rationale for study design, doses and control groups

eventual clinical interpretation of the study data and conclusions will be enhanced Overall strategic purpose of CSP Section 1.2: To confirm appropriateness of study design to fully address study objectives, so that credibility of

| | Regulatory representative | Biostatistics<br>representative | Physician representative |
|---|---|---|---|
| Does this section highlight and adequately address any potential limitations with study design (including study duration, blinding, choice of comparator, choice of dose, frequency of dosing and time of day, route of administration) that could be questioned by a Health Authority Reviewer? | Have current regulatory guidelines and any outstanding Health Authority concerns been addressed? | Has satisfactory justification been provided for key statistical design decisions (including study duration, blinding, choice of comparator, choice of dose, frequency of dosing and time of day, route of administration) and for any lack of concordance with standard research practices or medical/statistical/regulatory guidelines? | Has satisfactory medical and scientific justification been provided for key design decisions (including study duration, blinding, choice of comparator, choice of dose, frequency of dosing and time of day, route of administration) and for any lack of concordance with standard research practices or medical/statistical/regulatory guidelines? |

## Overall rationale and study population:

interviewing intervention delivered telephonically by pharmacists compared with usual care. disease, we will examine the impact of combining a shared decision making and behavioral After study completion, as a secondary aim, we will also use advanced predictive analytics to In this study of patients using at least one oral hypoglycemic therapy with poorly controlled

other generalized audiences about who is most likely to benefit from these patient engagement such as sociodemographic, clinical, medication use, and other motivational characteristics. examine whether patient response could have been predicted based on patient characteristics, techniques in real-world practice and target patients accordingly. intervention will provide policy-relevant information not only to Horizon BCBSNJ but also to This study and the use of predictive analytics to identify patients who most benefited from the

group. These eligibility criteria are described in further detail in Section 3. Seven-hundred patients who meet eligibility criteria will be allocated to the intervention

patient populations to a number of large insurers, including Horizon BCBSNJ. telephonic disease management services. The intervention will be delivered by trained and licensed pharmacists from a drug benefit management company that provides pharmacist-delivered has provided patient care services for other

The intervention is described in detail below.

# Intervention: Shared decision-making/Brief negotiated interviewing

decision-making tool and other patient materials in accordance with guidelines on conducting shared-decision making in practice.<sup>8,17</sup> solicit direct feedback. This patient feedback will be used to refine both the shared regular diabetic support groups and has received their commitment to participate and validated. 7,8,17,18 An online format for the decision aid will also be made available for of decision aid design and be based upon other decision aids that have been previously used to enhance interventional efforts. This decision aid will be developed using principles and pillbox that will prime them for telephonic encounters with pharmacists and will be volunteers. The study team has established a relationship with local providers who lead feedback on the decision aid and patient-oriented materials from a cohort of patient patient convenience. Prior to study launch, the study team will solicit direct patient Eligible patients will first be sent an invitation letter. This letter will include a decision aid

quickly and directly, an Interactive Voice Response System (IVRS) may also be used. One practices and Horizon BCBSNJ to help manage their patients. advantage of an IVRS is that it would provide a triage format for patients to contact the pharmacists directly after receiving the initial mailing. IVRS is frequently used in clinical To engage patients after the initial mailing and connect them with pharmacists more

driving a consensus of decision choices. For these encounters, the pharmacist will consist of a 2-stage process of identifying patients' motivations and participate by providing consent, the first telephonic encounter with the clinical to participate in the intervention and provide verbal informed consent. After agreeing to intervention group at least 4 times for the initial conversation. Each patient will be asked discussions about diabetes treatment options, goals and preferences, medication intervention and follow-up 'booster' phone calls. These telephonic encounters will include will use a semi-structured call guide developed by the study team for both the initial After the initial mailings, the pharmacists will attempt to reach each patient in the pharmacists

adherence, strategies for reducing barriers to adherence, implementing lifestyle not be contacted further. provided to encourage medication adherence. If patients do not provide consent, they will consultations, both discrete decision support and ongoing motivational support will be modifications and the benefits of maintaining blood glucose control. In these

guide that flows through the following phases (as part of the 2-stage process): In brief, the telephonic discussions with pharmacists will follow a semi-structured call

- (a) confirm treatment regimens,
- (b) discuss treatment goals and preferences,
- engage the patient in sharing potential medication non-adherence issues or lifestyle factors that may be contributing to poor control,
- (d) discuss potential barriers and willingness/readiness to modify behaviors, and
- engage the patient in identifying and agreeing upon a possible shared plan of modifications. behavioral strategies to improve glucose control and potential treatment

The two stages of the call guide are summarized, as follows:

- barriers to glucose control will be identified and discussed. consists of the shared decision-making process whereby discussions of issues and Stage 1 Shared-Decision Making: The first stage of the intervention encounter
- beliefs and concerns that may affect glucose control. the patients to elaborate and problem solve as well as illuminate underlying These discussions will occur in an open-ended manner, which will allow
- 0 adherence and treatment intensification to improve their disease control. and reconcile the relative personal risks and benefits of medication employed to aid in this encounter, which will to help the patient understand The previously-mailed decision aid developed for telephonic use will be
- 0 making process is patient involvement in the conversation and their care. self-report) or changing their medication adherence behaviors. who are already adherent to their current regimen (as determined by patient The shared decisions may involve intensification of therapies for patients Ultimately, the goal of this first stage of the shared-decision engagement
- about how to improve the patient's diabetes control, the second stage may involve adherence improvement as a goal. a behavioral interviewing engagement technique if the shared decision involves Stage 2: Once coming to a shared decision between the pharmacist and patient
- readiness for change. 19,20 using the Brief Negotiated Interview (BNI). This type of interviewing is identifying patients' readiness for change and level of behavior change posits that individuals move through a series of stages as they change built upon Prochaska's transtheoretical model of behavioral change, which This model incorporates an active listening model of counseling, behavior and identify interventions that are based on the individual's

- motivational enhancement techniques. short structured interview that incorporates brief feedback and advice with The BNI employs some features of motivational interviewing but through a
- 0 goals; (4) negotiating and advising. assessing readiness and developing discrepancy between behavior and support; (2) providing feedback; (3) enhancing motivation through The BNI proceeds through the following four main steps: (1) raising
- 0 intervention, there are established algorithms that will be used. To develop the structured BNI tool within the call guide for this
- The goal of this stage is to motivate patients to change behaviors

course of this intervention to adhere to their currently prescribed treatment, they are the patient's provider, either via letters, faxes, and phone calls, depending on urgency. side effect considerations, daily routines, any daily monitoring, and cost barriers. The modifications or issues with treatments, such as weight changes, low blood sugar, other shared plan may include medication non-adherence but potentially also lifestyle between the pharmacist and the patient. The barriers that will be addressed within the be identified, which will be modified upon each of the three subsequent encounters following treatment recommendations already set forth by their providers. performed by the patient's own treating physician. For patients who decide through the Ultimately any therapeutic decision (e.g. to change or intensify treatment) will be barriers and proposed plan for each patient will be communicated from the pharmacist to At the end of each conversation with the clinical pharmacist, a shared treatment plan will

and continue to engage the patient in discussions surrounding these topics. follow-up period. The follow-up "booster" phone calls will repeat some of these themes These pharmacist-delivered phone calls will occur a minimum of 4 times during the

# Primary and secondary outcome measures

centered medical homes and other population health programs. This laboratory information generalized estimating equations to compare changes. will be used to measure the change in HbA1c levels at the end of follow-up. We will use levels in each group. Horizon BCBSNJ receives laboratory information from over 200 patient-The primary outcome of interest will be the pre- to post-intervention change in mean HbA1c

measure, we will observe the mean PDC in each study arm and the proportion of patients medications will also be measured by pharmacy claims and their filling patterns. Adherence period. Other persistence measures including gaps in medication availability will also be achieving optimal adherence (defined by  $\geq$ 0.80 PDC) as adherence outcomes in the follow-up days that patients had medication available to them during follow-up. Using this PDC will be assessed using the proportion of days covered (PDC) measure, or the proportion of proportion of patients who achieved a HbA1c < 8.0%. Patients' adherence to their diabetes follow-up and the proportion of patients achieving optimal glycemic control, defined as the outcomes. The secondary glycemic outcomes will include mean HbA1c levels at the end of Secondary outcomes of interest include both glycemic outcomes and medication adherence

descriptively measured. More detail on the measurement is provided in Section 8.1. will be assessed using linear regression. Dichotomous outcomes will be compared using logistic regression, and continuous outcomes

#### Study duration

700 intervention patients will be identified and then followed for 12 months.

assessed using model discrimination and performance measures, including logistic regression, boosted regression and machine learning approaches.<sup>21-23</sup> delivered telephonic intervention. In brief, these predictive ability of these models will be adherence, other self-reported motivational characteristics, and receipt of the pharmacistpredicted based on patient factors, such as sociodemographic, clinical, medication use and examine whether the glucose control and medication adherence outcomes could have been After the completion of the study and database lock, we will use predictive analytics to

A schematic of the study design and duration are shown in Figure 1 below.

Figure 1. Schematic of the study design and patient identification and follow-up periods



# 1.3 Benefit/risk and ethical assessment

# Overall strategic purpose of CSP Section 1.3:

recent evaluation of product benefit/risk, and that the study is ethically defensible To ensure the benefits and risks of the study are complete, accurate and consistent with the most

| | | representative | Physician |
|---|---|---|---|
| Is the study defensible from an ethical standpoint? | benefit/risk? | representative complete, accurate and consistent with the most recent evaluation of the product's | Through consultation with the Global Safety Physician, is the stated benefit/risk |

intervention and control patients. In addition, we will seek study including have previously received approval for other studies using a similar study design and approach review board approval for this strategy after study protocol approval by AstraZeneca. We We have received Horizon Blue Cross Blue Shield Privacy Board approval to conduct this use of a HIPAA limited dataset to conduct analysis on all identified institutional

minimal, because healthcare data collected for the study were generated as part of routine overseen by the patient's provider. medication prescription data. In addition, all treatment decisions will ultimately be made and care, including clinical diagnoses of diabetes as well as relevant laboratory results and investigational products are being studied. Secondly, the risk to patients is no more than The risks to participating in this study are no more than minimal. First, no unapproved

and ages but no other identifying information. Limited information required for clinical care, identifiers and the medical record number will remain at Horizon in a password-protected file risk, only the minimum amount of data necessary will be shared, and the key between the Therefore, the primary risk to patients will be privacy of health information. To mitigate this access and access this information at any given time. In addition, all team members at both similar to other interventions already with Horizon, will be shared with and investigators will only have access to a HIPAA-limited dataset that includes dates and only a limited set of individuals directly caring for the patients will have have received appropriate and extensive training in data privacy.

#### 1.4 Study Design

The overall study design and flowchart for ENGAGE-DM is shown in Figure 2.

Figure 2

ENGAGE-DM Study Flowchart

STAGE

PROCESS



### 2. STUDY OBJECTIVES

| Control of the Contro | |
|---|---|
| Assuming favourable study outcomes, will the study objectives support worldwide Health Authority approval of the proposed indication and recommendations for use contained in the proposed CDS? | Regulatory representative |
| From a statistical point of view, are the study objectives clearly written and strictly focused on what questions the study should provide answers to in order to support the tollgate decision, proposed CDS and/or TPP/TPCs? | Biostatistics representative |
| From a medical and scientific point of view, are the study objectives clearly written and strictly focused on what questions the study should provide answers to in order to support the tollgate decision, proposed CDS and/or TPP/TPCs? | Physician representative |
| Overall strategic purpose of CSP Section 2: To ensure the objectives are aligned with the purpose of the study, so that the study will generate the right type of evidence needed to fully support its purpose in the clinical programme. | Overall strate To ensure the right type of e |

#### 2.1 Primary objective

| Primary Objective: | Outcome Measure: |
|---|---|
| To examine whether a two-stage process of | Glycosylated hemoglobin (HbA1c): |
| shared decision-making and behavioral | - Primary outcome: Pre- to post-intervention |
| interviewing improves glycosylated | change in mean HbA1c levels |
| hemoglobin (HbA1c) control and medication | - Mean levels in each study arm in the follow- |
| controlled diabetes | up period |
| | - Proportion of patients in each study arm |
| | follow-up period |
| | Medication adherence: |
| | - Continuous proportion of Days Covered |
| | period |
| | <ul> <li>Proportion of patients in each study arm<br/>achieving optimal adherence (PDC ≥0.80) in</li> </ul> |
| | the follow-up period |

### 2.2 Secondary objectives

| Secondary Objective: | Outcome Measure: |
|---|---|
| To develop prediction models and examine | Predictive statistics: |
| their ability to predict response to the study intervention based on baseline patient | <ul> <li>Cross-validated C-statistics (discriminative<br/>ability of the model)</li> </ul> |
| clinical, and medication use characteristics, as well as initial receptiveness to changing health behaviors | <ul> <li>Cross-validated R-squares (explained variation in treatment response)</li> </ul> |

#### 2.3 Safety objectives

| N/A | Safety Objective: |
|-----|-------------------|
| N/A | Outcome Measure : |

### 2.4 Exploratory objectives

| Exploratory Objective: Outcor | outcome Measure : |
|-------------------------------|-------------------|
| N/A N/A | |

#### S DISCONTINUATION AND WITHDRAWAL SUBJECT SELECTION, ENROLMENT, RESTRICTIONS,

# Overall strategic purpose of CSP Section 3:

subgroups). To define, and confirm appropriateness of, the study population, so that the proposed CDS will be fully supported by data obtained from the intended target population (including all relevant

| do they take into account the known safety profiles and restrictions of the investigational and comparator drugs? | do they investig |
|---|---|
| | Is the study population too refined because of unduly excluding or screening out too many subjects from the study? |

## Overall strategic purpose of CSP Section 3:

subgroups). fully supported by data obtained from the intended target population (including all relevant To define, and confirm appropriateness of, the study population, so that the proposed CDS will be

| Regulatory<br>representative | | | | representative | Biostatistics |
|---|---|---|---|---|---|
| Is the study population representative of the intended target population, taking into account restrictions required in terms of available safety data (e.g., use in women of childbearing potential), and if not what could be the possible consequences for the proposed CDS? | Has satisfactory justification been provided for any discrepancies between the study population and the intended target population – noting possible consequences for the proposed CDS? | Is the study population too refined because of unduly excluding or screening out too many subjects from the study? | do they take into account the known safety profiles and restrictions of the investigational and comparator drugs? | characteristics of the intended target population – noting any co-morbidities – and | From a statistical point of view, do the proposed entry criteria accurately define the |

consent will be obtained from patients allocated to the intervention group prior to participating commercially-insured population, so there should be no contamination for this study. in the intervention. Horizon BCBSNJ currently has no direct outreach to patients in this Each subject will meet all of the inclusion and exclusion criteria for this study. Informed

refined inclusion and exclusion criteria to existing administrative claims data. request and pulls the data. To identify study patients, Horizon analytics will first apply the is and what fields of information they may need for the pull. An analyst is then assigned to the Horizon has an analytics request database in house where they describe what the data request

In addition, we have previously received IRB approval at similar design and approach.<sup>24,25</sup> We have received Horizon Privacy Board approval for the design and approach in this study. for other studies using a

#### 3.1 Inclusion criteria

intervention and the validity of medication adherence measures, we will include patients in the members to enhance generalizability of the study population. Given the nature of the health management programs that collaborate with Horizon BCBSNJ but also include other approximately two hundred Patient-Centered Medical Homes (PCMHs) and other population capture of information. We plan to primarily include participants who receive care in patients who have Horizon BCBSNJ medical/prescription drug benefits ensures complete currently does not have any direct outreach efforts to patients in this population. Limiting to 1). First, commercially-insured beneficiaries will be chosen because Horizon BCBSNJ appropriate patients are included, while also maximizing generalizability of the study (Table The following inclusion criteria will be used to refine the study population to ensure

numbers to Horizon; however, initial feasibility estimates indicate that this is most of their intervention, we will only include patients in the study who have provided non-missing phone will be used to identify study patients, because multiple clinical guidelines concur that HbA1c study who are using at least one oral hypoglycemic medication (Table 2). A HbA1c of ≥8% patients (85%). levels this high indicate poor diabetes control. Lastly, due to the nature of the telephonic

Table 1. Patient inclusion criteria

| Criterion | Operationalization |
|---|---|
| Commercially-insured | Horizon BCBSNJ beneficiaries with PCP |
| beneficiaries | |
| Aged ≥18 years | Based on age on index date (the date of identification) |
| Receive all medical/prescription | Based on having data available on the index date (the date of |
| drug benefits through Horizon | identification) |
| On ≥1 one oral hypoglycemic | Filled ≥1 oral hypoglycemic agent within the 365 days prior the |
| agent | index date (the date of identification) in pharmacy claims |
| Latest HbA1c measurement ≥ | Have an HbA1c $\geq$ 8% within the 180 days prior to the index date |
| 8% (within previous 6 months) | (the date of identification) in laboratory claims |
| Provided phone number to | Based on Horizon BCBSNJ enrollment data |
| Horizon | |

Table 2. List of hypoglycemic agents for inclusion

| | : | | | | | : | 1 |
|---|---|---|---|---|---|---|---|
| Chlorpropamide Repaglinide Metformin Rosiglitazone Acarbose | aglinide | Metformin | Rosiglitazone | | Canagliflozin Sitagliptin Exenatide | Sitagliptin | Exenatide |
| | d | | c | | ( | ( | |
| Tolbutamide Nate | Nateolinide | | Pinglitazone | Miglital | Danaoliffozin Saxaolintin Liraolutide | Saxaglintin | Liraglutide |
| | ( | - | | | , | 1 | |
| Tolazamide | | **** | Troglitazone | | Empagliflozin Linagliptin Albiglutide | Linagliptin | Albiglutide |
| CONTRACTOR | | | ( | | , | , | , |
| Gliclazide | | | Tolazamide | | | Alogliptin Dulaglutide | Dulaglutide |
| : | | | E | | | | |
| Glipizide | | , | | | | | |
| ) | | | | | | | |
| Glyburide | | | | | | | |
| Glibencalamide | | | | | | | |
| Glimeniride | | | | | | | |
| Cimino | | | | | | | |

Fixed-dose combination products of these agents will also be included Note: GLP1 medications will also be measured, but patients will have to be on at least one other oral agent.

#### 3.2 Exclusion criteria

initial identification are using any insulin products. In specific, the management, measurement real-world nature of the study (Table 3). Because oral anti-insulin hypoglycemic agents are of medication adherence and use of patient engagement techniques in patients would differ if the primary medications of interest in this study, we will exclude patients who at the time of they are already using any human insulin or insulin analog A limited set of exclusion criteria will be used to identify eligible study patients to mimic the

Edition? Clinical Study Protocol Drug Substance NA Study Code D1843R00254

Table 3. Patient exclusion criterion

| Criterion | Operationalization |
|---|---|
| Currently using any insulin (listed below) | Insulin fill in previous 3 months in pharmacy claims data |

# List of insulin products for exclusion (any of the following - based on generic name)

- Rapid-acting: Lispro (Humalog), Aspart (Novolog), Glulisine (Apidra Short-acting: Regular (Humulin, Novolin, Velosulin)
- Intermediate-acting: NPH
- Long-acting: Glargine (Lantus), Detemir (Levemir)
- Mixes (Humulin, Novolin, Novolog, Humalog)

#### Subject enrollment

allocated to be eligible to receive the intervention. Patients allocated to the intervention group patients will not be contacted. also be identified by Horizon Analytics as a control group for analyses purposes only; these for auditing should re-confirmation of verbal consent be required. Seven hundred patients will pharmacist in consent to participate in the intervention. Verbal consent will be documented by the clinical will be contacted by phone by Patients will be identified by Horizon Analytics for the study. Seven hundred patients will be medical record. In addition, all calls will be recorded and available pharmacists and will be asked to provide informed

### Criteria for withdrawal

and the pharmacists will then no longer try to make contact with these patients. These strategies have been used in previous studies.<sup>26-29</sup> group will always have the option to withdraw their consent to participate in the intervention, determined by the Horizon Privacy Board. In addition, patients identified for the intervention BCBSNJ plan, but their data will be collected until the loss of continuous enrollment, as was Patients will not formally withdraw from the study unless they disenroll from a Horizon

# Withdrawal of the informed consent

own treating physician. Patients can choose to no longer participate in speaking with the therapeutic decision (e.g. to change or intensify treatment) will be performed by the patient's clinical pharmacists and withdraw their informed consent to participate in the study at any The intervention itself involves helping patients set health-related goals and ultimately any

# Discontinuation of the study

later not engage with the pharmacists during follow-up will not be further contacted Patients in the intervention arm who choose to not engage with the pharmacists or choose to

# STUDY PLAN AND TIMING OF PROCEDURES

outside of routine care. We will not be requiring patients to seek care at any specified intervals to obtain study data to mimic real-world clinical practice. There are no formal visits in this study or any clinical procedures that will be conducted

The study plan and timing of the study interventions are shown in Table 4 below.

Table 4. Timing of study interventions

| Study Arm | Initial<br>mailing | Initial call Follow-up call (#1) | | Follow-up<br>call (#2) | Follow-up<br>call (#3) |
|---|---|---|---|---|---|
| Intervention | Invitation | Consent + | Booster: | Booster: | Booster: |
| group | letter | Introduction | SDM + BNI | Introduction SDM + BNI SDM + BNI SDM + BNI | SDM + BNI |
| | | + SDM + | | | |
| | | BNI | | | 18/2018 |

# 4.1 Enrollment/screening period

the secondary predictive modelling study to identify the types of patients who will benefit within these conversations in a less structured or validated manner), but will also be tested in information that is relevant to the two patient engagement techniques (and could be captured The answers to these questions will not only help provide the pharmacists with additional call, these questions will be built into the semi-structured call guide used by the pharmacists. Patient Health Questionnaire-2 (PHQ-2)<sup>32</sup>. Administered towards the beginning of the initial marker for patient activation, and information about any baseline depression, including the readiness to change<sup>19</sup>, patient engagement, the Consumer Health Activation Index (CHAI), a self-reported medication adherence, such as the 1-item Morisky adherence question 30,31 survey questions. These additional items are anticipated to include a limited set of items on during the initial call after obtaining consent. These patients will be asked to respond to a few will capture some additional baseline information on patients assigned to the intervention arm To enhance the secondary predictive analytics aim of the study, from this intervention.

#### 4.2 Treatment period

intervention group will be contacted within their first month after identification, initially by mailed communication and then via the telephonic intervention. Follow-up "booster" telephonic phone calls by clinical pharmacists will be used at least 3 more times to support the Patients will be followed from the identification until the end of the study. Patients in the

#### 4.3 Follow-up period

As previously described, the follow up period will last for 12 months

## 5. STUDY ASSESSMENTS

### 5.1 Efficacy assessments

will use generalized estimating equations to compare the changes between the two groups. information will be used to measure the change in HbA1c levels at the end of follow-up. We levels to the end of follow-up. Horizon BCBSNJ receives laboratory information from over 200 patient-centered medical homes and other population health programs. This laboratory The primary outcome of interest will be the pre- to post-intervention change in mean HbA1c

descriptively measured. More detail on the measurement is provided in Section 8.1. period. Other persistence measures including and gaps in medication availability will also be achieving optimal adherence (defined by  $\geq$ 0.80 PDC) as adherence outcomes in the follow-up measure, we will observe the mean PDC in each study arm and the proportion of patients days that patients had medication available to them during follow-up. Using this PDC will be assessed using the proportion of days covered (PDC) measure, or the proportion of medications will also be measured by pharmacy claims and their filling patterns. Adherence proportion of patients who achieved a HbA1c <8.0%. Patients' adherence to their diabetes outcomes. The secondary glycemic outcomes will include mean HbA1c levels at the end of be assessed using linear regression. follow-up and the proportion of patients achieving optimal glycemic control, defined as the Secondary outcomes of interest include both glycemic outcomes and medication adherence Dichotomous outcomes will compared using logistic regression, and continuous outcomes will

#### 5.2 Safety assessments

N/A

#### 5.3 Other assessments

N/A

#### 5.4 Pharmacokinetics

N/A

### 5.5 Pharmacodynamics

N/A

#### 5.6 Biomarker analysis

N/A

## 9 SAFETY REPORTING AND MEDICAL MANAGEMENT

become aware of any adverse event in a patient with an AstraZeneca product, they will report There are no investigational products being examined in this study. If the clinical pharmacists

Clinical Study Protocol
Drug Substance NA
Study Code D1843R00254
Edition<sup>2</sup>
Date

and/or manufacturer) through the spontaneous adverse event reporting system (Website: aware of any adverse event that are associated with manufacturers other than AstraZeneca, any adverse event to AstraZeneca, refer to section 6.4. In addition, the clinical pharmacist is is involved in an observational study in which no study medications are administered subjects/health care providers who report the adverse events (AEs) to disclose that the subject http://www.fda.gov/safety/medwatch/howtoreport/ucm053087.htm. We may request the study http://www.fda.gov/Drugs/GuidanceComplianceRegulatoryInformation/Surveillance/Adverse they will be encouraged to report them according to local requirements (health authority DrugEffects/ucm115894.htm). For serious adverse events (SAE), please refer to FDA website

# 6.1 Definition of adverse events

abnormal results of an investigation (e.g., laboratory findings, electrocardiogram). In clinical of a pre-existing medical condition following or during exposure to a pharmaceutical product, run-in or washout periods, even if no study treatment has been administered studies, an AE can include an undesirable medical condition occurring at any time, including can be symptoms (e.g., nausea, chest pain), signs (e.g., tachycardia, enlarged liver) or the whether or not considered causally related to the product. An undesirable medical condition An adverse event is the development of an undesirable medical condition or the deterioration

The term AE is used to include both serious and non-serious AEs

# 6.2 Definitions of serious adverse event

the following criteria: A serious adverse event is an AE occurring during any study phase that fulfills one or more of

- Results in death
- Is immediately life-threatening
- Requires in-patient hospitalisation or prolongation of existing hospitalisation
- ability to conduct normal life functions Results in persistent or significant disability/incapacity or substantial disruption of the
- Is a congenital abnormality or birth defect
- intervention to prevent one of the outcomes listed above Is an important medical event that may jeopardise the subject or may require medical

# 6.3 Recording of adverse events

# 6.3.1 Time period for collection of adverse events

completion of the study. Adverse events will be collected from time of signature of informed consent throughout the

need to report it to AZ as indicated in Section 6.4. the clinical pharmacists identify any adverse event with an AstraZeneca product they will course of regular clinical care because there are no investigational products being studied. If As previously described, any adverse events from the medications will be handled during the

# Reporting of adverse events and serious adverse events

is preferred method). to AstraZeneca's designated mailbox send the SAE report and accompanying cover page by way of fax to AstraZeneca's designated If the clinical pharmacist becomes aware of an AE or an SAE with an AZ product they need to or send SAE report and accompanying cover page by way of email (email

#### 6.4.1 Reporting timelines

relevant follow-up information is also provided to AstraZeneca within one day of initial initial reporting, to the AZ representative. If a non-serious AE becomes serious, this and other corrections to data previously submitted on SAEs, within the same timelines specified for with AZ products. The clinical pharmacist will also report all follow-up information or and life-threatening cases and within five calendar days of initial receipt for all other SAEs Safety Data Entry Site receives a report within one calendar day of initial receipt for all fatal clinical pharmacist to compile all necessary information and ensures that the AZ Patient AZ representative (e.g. Patient Safety personnel at Marketing Company) will work with the receipt as described above. When informed by the clinical pharmacist that a SAE has occurred with an AZ product, the

#### 6.4.2 Variables

The following variables will be collected for each adverse event with an AZ product;

- Adverse event (verbatim)
- The date when the adverse event started and stopped
- Maximum intensity
- Whether the adverse event is serious or not
- Investigator causality rating against the Investigational Product (yes or no)
- Action taken with regard to the AZ medication
- Whether the adverse event caused patient's withdrawal from study (yes or no) and
- Outcome

In addition, the following variables will be collected for SAEs:

Date adverse event met criteria for an SAE

- Date Investigator became aware of an SAE
- Adverse event is serious due to
- Date of hospitalization
- Date of discharge
- In case of fatal reports:
- Probable cause of death,
- Date of death,
- Autopsy performed,
- Causality assessment in relation to study procedure(s), and
- Description of adverse event.

shown in Section 6.2. On the other hand, a stroke that results in only a limited degree of several hours may be considered severe nausea, but not an SAE unless it meets the criteria intensity need not necessarily be considered serious. For example, nausea that persists for shown in Section 6.2 disability may be considered a mild stroke but would be an SAE when it satisfies the criteria intensity whereas seriousness is defined by the criteria in Section 1.2. An AE of severe It is important to distinguish between serious and severe AEs. Severity is a measure of

#### 6.5 Overdose

that specified in the US Prescribing Information unless otherwise prescribed by the physician An overdose is defined as a subject receiving a dose of an AstraZeneca product in excess of

Overdose in itself is not considered to be an AE or SAE.

must inform appropriate AZ representatives immediately, or no later than 24 hours of when he If an overdose on an AZ product occurs in the course of the study, then the clinical pharmacist or she becomes aware of it.

apply. For other overdoses, reporting must occur within 30 days For overdoses associated with a SAE with an AZ product, the standard reporting timelines

Form can be provided upon request): The following information should be provided in the event of an Overdose (Overdose Report

Details of the Patient who was dispensed the AZ drug (Patient Identification number)

- study participant?) Details of the Patient who took the overdose (demographic information, was patient a
- stop dates) Details of the drug overdose (total daily dose, route, formulation, Overdose start and
- Was the overdose accidental or intentional?
- Was the overdose associated with an adverse event (serious or non-serious)
- indicate if the event is ongoing Provide an Adverse Event description. Provide start and stop dates of the event, or
- Provide the Clinical Pharmacist's signature and date.

#### 6.6 Pregnancy

study, the clinical pharmacist will request that the patient to seek advice from the patient's and any other relevant medical measures. whether the patient is still appropriate for continuation on the medication during pregnancy care physician on whether the potential benefit justifies the potential risk to the fetus, and If the clinical pharmacist is aware of a patient who becomes pregnant during the course of the

their outcomes in accordance with the standard clinical study protocol instructions are responsible for recording and reporting pregnancies for patients using AZ products and Pregnancy in itself is not considered to be an AE or SAE. However, the clinical pharmacist

#### 6.6.1 Maternal Exposure

whether the patient is still appropriate for continuation during pregnancy and any other care physician on whether the potential benefit justifies the potential risk to the fetus, and study, the clinical pharmacist will request that the patient to seek advice from the patient's If the clinical pharmacist is aware of a patient who becomes pregnant during the course of the relevant medical measures.

of all pregnancies (spontaneous miscarriage, elective termination, ectopic pregnancy, normal SAEs. Elective abortions without complications should not be handled as AEs. The outcome abnormalities/birth defects and spontaneous miscarriages should be reported and handled as drug may have interfered with the effectiveness of a contraceptive medication. Congenital Pregnancy itself is not regarded as an adverse event unless there is a suspicion that the AZ documented birth or congenital abnormality) while using any AZ product should be followed up and

later than 24 hours of when he or she becomes aware of it. informs the appropriate AstraZeneca representatives within 1 day i.e., immediately but no If any pregnancy occurs in the course of the study while using an AZ product, then the clinical

pregnancies. SAEs (see <<Section: Reporting of serious adverse events>>) and within 30 days for all other information is provided to the AZ Patient Safety data entry site within 1 or 5 calendar days for The designated AZ representative works with the clinical pharmacist to ensure that all relevant

The same timelines apply when outcome information is available

#### 6.6.2 Paternal Exposure

and reported in accordance with the processes written in Section 6.6.1. information and follow-up on the pregnancy. The outcome of the pregnancy is also followed exposure. The female partner of the patient will be asked to consent to allow collection of then the clinical pharmacist should inform AZ within the same timeframe as the maternal If paternal exposure pregnancy occurs in the course of the study while using an AZ product,

# 6.7 Management of IP related toxicities

N/A

# 6.8 Study governance and oversight

study team is not necessary. Due to the low-risk nature of this study, a data safety monitoring committee outside of the

# 7 INVESTIGATIONAL PRODUCT AND OTHER TREATMENTS

N/A

# 8. STATISTICAL ANALYSES

# Overall strategic purpose of CSP Section 8:

clinical interpretation of the study data and conclusions will be enhanced. To confirm appropriateness of statistical methodology and assumptions, so that credibility of eventual

| Physician | From a medical point of view, does the statistical approach address all the study |
|---|---|
| representative | objectives and will the analyses likely result in clinically meaningful and interpretable data to support the tollgate decision, proposed CDS and or TPP/TPCs: |
| | Has a robust clinical and statistical justification been provided for any non- |
| | inferiority/equivalence margins? |

| } | V |
|---|---------------------------------------------|
| 5 | erall |
| • | stra |
| | Overall strategic purpose of CSP Section 8: |
| • | [mg |
| | pose |
| , | of |
| | CSP |
| • | Sec |
| • | tion |
| | 8: |
| - | |

clinical interpretation of the study data and conclusions will be enhanced. To confirm appropriateness of statistical methodology and assumptions, so that credibility of eventual

| | Regulatory representative | | | Biostatistics<br>representative |
|---|---|---|---|---|
| Does this section highlight and adequately justify any lack of concordance with such guidelines and advice (noting any potential consequences for the proposed CDS)? | Is the statistical approach in agreement with current regulatory guidelines and any outstanding Health Authority statistical concerns? | Could an independent statistician replicate the analyses? | Has satisfactory statistical justification been provided for the choice of analysis methods (including any interim analyses), definition of analysis sets and calculations of sample size (including statistical and clinical justification for any non-inferiority/equivalence margins)? | Does the statistical approach address all the study objectives and will the analyses likely result in clinically meaningful and interpretable data to support the tollgate decision, proposed CDS and or TPP/TPCs? |

Statistical analyses will be conducted by the study team at with input and review from the fully study team, including AstraZeneca and Horizon BCBSNJ

### 8.1 Statistical considerations

#### Aim 1 (Primary Objective):

conducted among patients who provided informed consent versus the control group. carefully matched using observable covariates. Secondary analyses for all outcomes will be by comparing only consenting patients to the identified controls, even if patients were an intention-to-treat basis. This approach will minimize the potential selection bias introduced be conducted among all patients identified for the control group and the intervention group on HIPAA limited dataset on all patients for the purpose of analysis. The primary analyses will We have received Horizon Blue Cross Blue Shield Privacy Board approval to receive a

groups. Any observed imbalance between the groups will be controlled for using multivariable will use generalized estimating equations to compare the changes between the two study meaningful differences in these levels within the 11 to 12-month follow-up period. 24,25 follow-up. Because the primary outcome is HbA1c change, we expect to see clinically 200 patient-centered medical homes and other population health programs and other practices levels to the end of follow-up. Horizon BCBSNJ receives laboratory information from over regression. This laboratory information will be used to measure the change in HbA1c levels at the end of The primary outcome of interest will be the pre- to post-intervention change in mean HbA1c

(PDC), by dividing the number of days with medication available by the number of days during follow-up.<sup>33</sup> Using this PDC measure, we will observe the mean PDC in each study of days that patients had medications available to them, or the proportion of days covered considered to be interchangeable. From these supply diaries, we will calculate the proportion early or overlapping fills can accumulate up to 180 days of excess supply in the supply diary. observed fills after initiation based on dispensing date and days' supply. The supply for any their filling patterns. For each medication, we will create a drug supply diary linking all Patients' adherence to their diabetes medications will be measured by pharmacy claims and major quality measures used to assess the performance of health plans, including HEDIS proportion of patients who achieved a HbA1c <8.0%, which is the threshold for the most outcomes. The secondary glycemic outcomes will include mean HbA1c levels at the end of adherence outcomes in the follow-up period. group and the proportion of patients achieving optimal adherence (defined by  $\geq 0.80$  PDC) as Different drugs in the same chemically-related therapeutic class (e.g., sulfonylureas) will be follow-up and the proportion of patients achieving optimal glycemic control, defined as the Secondary outcomes of interest include both glycemic outcomes and medication adherence

censored on that date, and the PDC will be calculated based on the number of days available. intensify therapy (e.g., adding a second oral diabetes medication or injectable medication). measurement even when patients switch (e.g., switch from metformin to a sulfonylurea) or they will considered to be adherent for that day. This definition allows for outcome In this PDC measurement, if patients had at least one antidiabetic medication available, then If a patient loses continuous eligibility during the year after the index date, they will be

study group. 24,34 augmentation, discontinuation and other changes in prescription patterns will also be ≥80% PDC), and gaps in medication availability. For these definitions, rates of switching, be measured. This approach to multiple medications has been used in other studies by our period. If insulin is used adjunctively or instead of oral therapy, persistence to insulin will also as a gap in supply of  $\geq$ 60 days following exhaustion of the drug supply in the follow-up period that medication was used for. Persistence to medications will also be assessed, defined adjusting the denominator for new medication based on the number of days in the follow-up measured descriptively. Adherence to each diabetes medication will be measured using PDC, individual anti-diabetic medication, the proportion of patients who were adherent (defined by Other medication adherence measurements will also be assessed, including adherence to each

#### Aim 2 (Secondary Objective):

PDC > 0.80). Specifically, we will evaluate prediction models with respect to their ability to characteristics predict glucose control (e.g., HbA1c<8%) and medication adherence (e.g., to this type of intervention. In this aim, we will retrospectively examine whether these telephonic intervention. The goal is also to identify patients who were most likely to respond medication use, and other motivational characteristics, and receipt of the pharmacist-delivered could have been predicted based on patient factors, such as sociodemographic, clinical, As a secondary aim, we will use predictive analytics to examine whether the clinical outcomes

and medication adherence targets during the follow-up period discriminate and explain variation between patients who did and did not meet the glycemic

the models will include only predictors available from administrative claims and not screening assessment during the initial pharmacist-delivered telephonic encounter. These demographic, clinical, and medication use characteristics and information from the brief and PDC and will include different numbers of predictor variables, in a method similar to payers alike. For these models, the outcome will be treatment response as defined by HbA1c adherence, respectively, and will be meaningful measures for providers, policymakers, and considered to be clinically meaningful cutpoints for achieving optimal control for diabetes and characteristics as predictors. We will model these particular outcomes because these are the survey, baseline adherence as measured by pharmacy claims, and response to the information from patient self-report. We will also assess the correlation between responses to Horizon BCBSNJ outpatient pharmaceutical, medical, and laboratory claims files. Some of baseline demographic, clinical, and medication use characteristics will be measured using previous work. 35,36 As predictors in these models, we will incorporate patients' baseline for patients in both the treatment and control groups, incorporating different patient (e.g., HbA1c<8% and PDC>0.80), we will develop and estimate a series of regression models To assess the ability to predict patients who will respond to the intervention, for each outcome

are any differences in predictive ability. estimation will be repeated among relevant patient subgroups (e.g., gender, age) to see if there which set of characteristics are most predictive of the response to the intervention. Model intervention patients who had at least 1 telephonic encounter with a pharmacist to examine receiving the intervention. We will also repeat the analyses among the subgroup of term so the logistic regression will provide estimates on all patients and not just those follow-up period.35 to assess the ability to predict medication adherence and glycemic control in the subsequent subsequent medication adherence, we will also include initial post-baseline filling information as initial filling information have been shown in previous work to be highly predictive of initial screening characteristics (e.g., Morisky score, PHQ-2 score, CHAI score). In addition, models that include these predictors as well as baseline medication adherence information and includes only demographic and clinical characteristics. We will then estimate additional For each outcome (e.g., HbA1c<8% and PDC>0.80), we will first estimate a model that Receipt of the pharmacist intervention will be tested using an interaction

similar likelihood of experiencing the clinical outcomes clustering patients who are most likely to respond will also explored, including machine approach is considered to be one of the best prediction approaches. Alternative methods of incorporate a number of non-linear associations between the predictors and the outcomes; this interactions among the predictors.<sup>37</sup> Through these many regression trees, the model can a prediction model through building many regression trees with the potential for many logistic regression and generalized boosting regression, a data mining technique that generates Models among each of the control and intervention groups will be predicted using both learning to develop models algorithmically, to partition patients into clusters that have a

degree of variation explained by the model, ranging from 0 (no variation explained) to 1.0 (all the C-statistic. A C-statistic of 1.0 indicates perfect prediction and a value of 0.5 indicates no of the model to distinguish between patients who do and do not experience the outcome, by validation results over the 10 repetitions.<sup>22</sup> different partitions (leaving 10% of the data out each time) 10 times and averages the will perform 10-fold cross-validation, which randomly partitions a sample of data into bias associated with evaluating prediction accuracy in the same data used for estimation, we linear regression, using R-squares to examine predictive ability. To avoid "over optimism" well as continuous PDC at the end of the follow-up period using linear regression and boosted variation explained) <sup>39</sup>. As secondary analyses, we will also model the change in HbA1c as association. 21,22 Pseudo R-squares will be used to assess model performance by examining the To compare the accuracy of the prediction models, we will compare discrimination, the ability

results to also be generalizable to other chronic disease medication management programs about how to manage their members who have poorly-controlled diabetes. We expect these will have specific ramifications for Horizon BCBSNJ as well as other payer organizations types of patients who may respond to these patient engagement techniques. These findings The results of these predictive analytic efforts will help inform payers and providers about the

#### 8.2 Sample size estimate

adherence outcomes (Table 6). including clustering and non-differential loss-to-follow up between the study groups (Table  $\alpha$ =0.05, 1- $\beta$ =0.80, A1c standard deviation=1.9, and a verbal informed consent rate of 45%, control group should be sufficient to detect an average change of 0.5% in A1c, assuming an We anticipate that identification of at least 700 individuals in the intervention group and . With this sample size, we should also have the ability to detect differences in the

observed in prior work with clinical pharmacists.8 This sample size would also provide 0.5% in the study population, these contacted patients must have a underlying mean A1c change of ~0.49% (Figure 3). This difference is in line with what clinical guidelines consider studies that have used a similar approach.<sup>25</sup> In order to observe an overall A1c difference of usable follow-up data. This proportion of reached patients has been observed in prior, pilot intervention group who are likely to be reached by pharmacists (45%), at least 236 will have study outcomes (glycemic control and medication adherence). enough patients for the predictive analytics work, given the relative non-rare nature of the to be a clinically meaningful difference in glycemic control. This A1c difference has been Based on feasibility information from Horizon, we anticipate that of the 315 patients in the

Table 5. Justification: A1c power calculation parameters and ranges

| Range of parameters: input ranges | A1c difference: 0.5% |
|---|---|
| | Sample size (N range)/group |
| A1c SD: $1.9> N_1$ | 228 |
| Intra-cluster correlation | 235 |
| $(N_2=N_1*1.03)$ | |
| Loss-to-follow-up (LTF): 15-30% (best case: 276, worst case: 335) | (best case: 276, worst case: 335) |
| The second secon | |

| | Total | $(N_4=N_3/rate)$ | Pharmacist contact rate: 35-50% | $(N_3=N_2/[1-rate])$ |
|---|---|---|---|---|
| 696 patients/arm | 45% reach rate and 25% LTF: | 1 | (best case: 552, worst case: 959) | |

Power  $(1-\beta)$ : 0.80; Alpha  $(\alpha)$ : 0.05

# Explanation of study parameters - Primary outcome (A1c)

- between the groups. This would be non-differential between study groups. average baseline A1c values. The most commonly cited value is 1.9, assuming equal variances 1) Standard deviation of A1c: ranges between 1.0 and 2.0, depending on study length and
- study groups. within PCP clinics (~0.03 for small pilot studies). This would be non-differential between 2) Intra-cluster correlation: Other studies have also incorporated intra-cluster correlation (ICC)
- end of the calendar year, we anticipate that there could be some non-differential loss-to-3) Loss-to-follow-up: Due to the potential for patients changing insurances particularly at the A1cs, despite restricting to patients whose providers have at-risk contracts with Horizon follow-up of patients in the study. There may also be patients who do not have follow-up
- reached by the pharmacists delivering the intervention. 4) Pharmacist contact rate: We anticipate that approximately 45% of the patients will be

Table 6. Justification: Adherence power calculation parameters and ranges

| Range of parameters: input ranges | Difference in mean PDC: 5% |
|-----------------------------------------|-----------------------------------|
| 1 | Sample size (N range)/group |
| Baseline adherence: 50%> N <sub>1</sub> | 253 |
| Intra-cluster correlation | 261 |
| $(N_2=N_1*1.03)$ | |
| Loss-to-follow-up (LTF): 10-25% | (best case: 290, worst case: 347) |
| $(N_3=N_2/[1-rate])$ | |
| Pharmacist contact rate: 35-50% | (best case: 580, worst case: 993) |
| $(N_4=N_3/rate)$ | |
| Total | 45% reach rate and 15% LTF: |
| | 682 patients/arm |

Power  $(1-\beta)$ : 0.80; Alpha  $(\alpha)$ : 0.05

# Explanation of additional study parameters - Secondary outcome (Adherence)

- 1) Baseline adherence:
- 5% absolute difference in mean PDC has been seen in previous intervention studies and is considered to be a clinically meaningful difference<sup>16,24</sup>
- Assuming ~50% baseline adherence based on previous literature<sup>24</sup>
- will be captured on all patients included in the study by definition, enabling the calculation of could be some non-differential loss-to-follow-up of patients in the study. Prescription claims adherence until loss of continuous eligibility. 2) Loss-to-follow-up: Due to the potential for patients changing insurances, we anticipate there

Figure 3. Schematic of analytic plan



## **8.3** Definitions of analysis sets

The full analysis set (Intention-to-Treat principle) will be used for the study analysis

# 8.4 Outcome measures for analyses

Please see Section 8.1 for further detail

# 8.5 Methods for statistical analyses

Please see Section 8.1 for further detail.

# 9. STUDY AND DATA MANAGEMENT

# 9.1 Training of study site personnel

all of these staff, and that any new information relevant to the performance of this study is staff involved in the study. The Principal Investigator will also train the clinical pharmacists at forwarded to the staff involved. The Principal Investigator will maintain a record of all study The Principal Investigator will ensure that appropriate training relevant to the study is given to in the conduct of the intervention, in accordance with the study timeline.

### 9.2 Monitoring of the study

investigators: During the study, an AstraZeneca representative will have regular contacts with the study

- Provide information and support to the Investigator(s)
- Confirm that the investigational team is adhering to the protocol

staff need information and advice about the study conduct. The AstraZeneca representative will be available as necessary if the Investigator(s) or other

#### 9.2.1 Source data

N/A

#### 9.2.2 Study agreements

ultimately be approved by patients' own prescribing physicians communicated with by the study pharmacists, and all treatment plans and changes will Clinical Study Protocol, or equivalent, for this study. Patients' physicians will be The Principal Investigator should comply with all the terms, conditions, and obligations of the

## 9.2.3 Archiving of study documents

The Investigator follows the principles outlined in the Clinical Study Protocol

### 9.2.4 Deviation from the clinical study protocol

medical reasons, or where the changes involve only logistical or administrative aspects of the or change is necessary to avoid an immediate hazard to the subjects or for other compelling clinical study (e.g., changes to the organisation/structure of the AstraZeneca, the approval based on its deliberations. However, this shall not apply to cases where the deviation documented agreement between the Principal Investigator and AstraZeneca or the IRB AstraZeneca, the job title of the Investigator, and monitors). name/department name of the study site, the address or phone number of the study site or The Investigator(s) must not deviate from or make any changes to the protocol without

# 9.3 Study timetable and end of study

will begin and end in Quarter 3 2016. The study is expected to start in Quarter 3 2016 and to end by Quarter 2 2017. Recruitment

#### Completion of the study

completion of the study to the IRB and AstraZeneca Upon terminating the study, the Principal Investigator/Investigator will report in writing the

# Data management by and Horizon Analytics

efforts). All data will be transferred by Horizon using a File Transfer Protocol (FTP) site from and download data to local, secure servers. designated person at each site will securely log in using a designated username and password Horizon in accordance with current practices. Horizon uploads PHI/data and only one the intervention (similar to data already shared with Information (PHI)/data to the study partners, mainly to the missing data. Horizon Analytics will disclose a very limited set of Protected Health Data management will be primarily performed by Horizon Analytics and secondarily by Data queries will be raised for inconsistent, impossible or for other Horizon outreach pharmacists to conduct

eligible patients. information, and laboratory information. This information will be necessary to intervene upon information, pharmacy contact information, primary care provider/practice, pharmacy claims the intervention and include the following information: demographic information, contact outreach interventions to Horizon members. The PHI/data will be the minimum necessary for These data will be similar to data that are routinely shared with The study patients will be identified by Horizon Analytics for already for other

information, laboratory information, and medical claims. This information will be necessary encrypted by a study key only known to Horizon, as follows: age, sex, pharmacy claims to assess the impact of the intervention. include a limited dataset that includes dates but no other identifying information, The PHI that will be disclosed by Horizon to the aforementioned study partners at the

environments so that privacy and security from unstructured data will be maintained. Data site from Horizon and unstructured, segmented ASCII datafiles to be maintained within in HIPAA privacy and security policies. All data will be transferred by Horizon using a FTP contain any individual PHI. The data files will remain on the secure server under password environments and files provided by Horizon will only be in aggregated form and will not the study. Additionally, all personnel with access to Horizon data will have had recent training maintained for the exact period necessary to conduct the work. protection and no datafiles will reside on local computers. In addition, access will only be will not leave the controlled server, and any information brought out of these secure files necessary. All data analysis will be performed within these traditional database traditional database/data warehouse environments (to The data will be stored on password-protected servers at each of the entities participating in in accordance with current practices for outreaches) using the minimum number of ) and Excel datafiles (to

responsibilities of the various functions and personnel involved in the data management and have been processed correctly. The Data Management Plan will also clarify the roles and procedures will be applied to each stage of data handling to ensure that all data are reliable The data will be validated as defined in the Data Management Plan. Quality control

revealing data may thereafter be added and the final database will be locked. When all data have been validated and locked, a clean file will be declared. Any treatment

### 10. ETHICAL AND REGULATORY REQUIREMENTS

# 10.1 Ethical conduct of the study

regulatory requirements and the AstraZeneca policy on Bioethics and Human Biological Declaration of Helsinki and are consistent with ICH/Good Clinical Practice, applicable The study will be performed in accordance with ethical principles that have their origin in the

### 10.2 Subject data protection

and control patients. The intervention itself poses no more than minimal risk because of the share a HIPAA limited dataset with decisions are also still being made by the patients' own physicians. extensive security and privacy measures undertaken by the study team; any treatment Horizon to share PHI with As previously described in Section 3.10, we have received a waiver of authorization for for the purpose of the intervention and for Horizon to to conduct analyses on all identified intervention

# 10.3 Ethics and regulatory review

these documents to the applicable IRB Committee, and to the study site staff. and/or materials to be provided to the subjects. The Investigator will ensure the distribution of An Institutional Review Board (IRB) from the will approve the final study protocol, including any other written information

required by local regulations, the protocol should be re-approved by the IRB Committee the written approval to AstraZeneca before enrollment of any subject into the study. If annually. The opinion of the IRB Committee should be given in writing. The Investigator should submit

#### 10.4 Informed consent

recorded and available for auditing intervention. All calls with patients, including those in which this consent is obtained, will be will obtain verbal informed consent from patients prior to administering the

# Changes to the protocol and informed consent form

Investigator and AstraZeneca. Study procedures will not be changed without the mutual agreement of the Principal

protocol (Revised Clinical Study Protocol). documented in a study protocol amendment and where required in a new version of the study If there are any substantial changes to the study protocol, then these changes will be

national regulatory authority approval, before implementation. Local requirements are to be followed for revised protocols. The amendment is to be approved by the relevant Ethics Committee and if applicable, also the

each Principal Investigator(s). For distribution to Ethics Committee see Section 10.3 AstraZeneca will distribute any subsequent amendments and new versions of the protocol to

by each Ethics Committee. If local regulations require, any administrative change will be communicated to or approved

### 10.6 Audits and inspections

related activities and documents, to determine whether these activities were conducted, and contacted by a regulatory agency about an inspection at the centre applicable regulatory requirements. The Investigator will contact AstraZeneca immediately if Practice (GCP), guidelines of the International Conference on Harmonisation (ICH), and any data were recorded, analysed, and accurately reported according to the protocol, Good Clinical purpose of an audit or inspection is to systematically and independently examine all studymay perform audits or inspections at the centre, including source data verification. Authorised representatives of AstraZeneca, a regulatory authority, or an Ethics Committee

## 11. LIST OF REFERENCES

- -Hogan P, Dall T, Nikolov P, American Diabetes A. Economic costs of diabetes in the US in 2002. *Diabetes care*. Mar 2003;26(3):917-932.
- 12 in urban African-Americans. IX. Provider adherence to management protocols el-Kebbi IM, Ziemer DC, Musey VC, Gallina DL, Bernard AM, Phillips LS. Diabetes Diabetes care. May 1997;20(5):698-703.
- S medicine. Aug 4 2005;353(5):487-497. Osterberg L, Blaschke T. Adherence to medication. The New England journal of
- 4 *Health Expectations.* 2006;9(1):25-36. between patients with chronic conditions and their clinicians: the case of diabetes Montori VM, Gafni A, Charles C. A shared treatment decision-making approach
- S encounters. Patient education and counseling. Mar 2006;60(3):301-312. Makoul G, Clayman ML. An integrative model of shared decision making in medical
- 6 what does it mean? (or it takes at least two to tango). Social science & medicine. Mar 1997;44(5):681-692. Charles C, Gafni A, Whelan T. Shared decision-making in the medical encounter:
- .7 2013;13:301. 2 diabetes: a randomized trial in primary care. BMC health services research Branda ME, LeBlanc A, Shah ND, et al. Shared decision making for patients with type
- $\infty$ screening decisions. The Cochrane database of systematic reviews. 2014;1:CD001431 Stacey D, Legare F, Col NF, et al. Decision aids for people facing health treatment or

- 9. primary care: the ASPIRE randomized clinical trial. Jama. Aug 6 2014;312(5):502-Saitz R, Palfai TP, Cheng DM, et al. Screening and brief intervention for drug use in
- 10. assessment of an intervention. AIDS patient care and STDs. Apr 2004;18(4):229-238. improve adherence to antiretroviral therapy: development and qualitative pilot Adamian MS, Golin CE, Shain LS, DeVellis B. Brief motivational interviewing to
- 1. young people. Drug and alcohol review. Dec 2003;22(4):391-399. model for public health purposes: a brief application of motivational interviewing with McCambridge J, Strang J. Development of a structured generic drug intervention
- 12. of substance abuse treatment. Jan 2013;44(1):139-142. based multicomponent intervention for smokers with substance use disorders. Journal Bernstein SL, Bijur P, Cooperman N, et al. Efficacy of an emergency department-
- 13 randomized controlled pilot feasibility trial. Patient preference and adherence. 2014;8:1555-1569. improve adherence to inhaled corticosteroids among adult asthmatics: results from a Lavoie KL, Moullec G, Lemiere C, et al. Efficacy of brief motivational interviewing to
- 14. Design of the OPTIMA Trial. Osteopor Int. 2010;21:137-144. Motivational Interviewing to Improve Adherence with Osteoporosis Medications: Solomon DH, Gleeson T, Iversen M, et al. A Blinded Randomized Controlled Trial of
- 15. 2011;82(1):117-122. American adolescents with asthma. Patient education and counseling. Jan interviewing intervention to promote medication adherence among inner-city, African-Riekert KA, Borrelli B, Bilderback A, Rand CS. The development of a motivational
- 16, review. Annals of internal medicine. Dec 4 2012;157(11):785-795 self-administered medications for chronic diseases in the United States: a systematic Viswanathan M, Golin CE, Jones CD, et al. Interventions to improve adherence to
- 17. 2009;169(17):1560-1568. decision aid: a randomized trial. Archives of internal medicine. Sep 28 Mullan RJ, Montori VM, Shah ND, et al. The diabetes mellitus medication choice
- 18 care. Jun 2010;48(6 Suppl):S153-158. comparative effectiveness into practice: the case of diabetes medications. Medical Shah ND, Mullan RJ, Breslin M, Yawn BP, Ting HH, Montori VM. Translating
- 19. behaviors. Progress in behavior modification. 1992;28:183-218. Prochaska JO, DiClemente CC. Stages of change in the modification of problem
- 20. Psychology, American Psychological Association. Jan 1994;13(1):39-46. Prochaska JO, Velicer WF, Rossi JS, et al. Stages of change and decisional balance for 12 problem behaviors. Health psychology: official journal of the Division of Health
- 21. prediction. Circulation. Feb 20 2007;115(7):928-935. Cook NR. Use and misuse of the receiver operating characteristic curve in risk
- 22 models: a framework for traditional and novel measures. Epidemiology. Jan Steyerberg EW, Vickers AJ, Cook NR, et al. Assessing the performance of prediction 2010;21(1):128-138
- 23 improvement calculations to measure usefulness of new biomarkers. Statistics in Pencina MJ, D'Agostino RB, Sr., Steyerberg EW. Extensions of net reclassification *medicine*. Jan 15 2011;30(1):11-21.

- 24. after Myocardial Infarction. The New England journal of medicine. 2011;365:2088-Choudhry NK, Avorn J, Glynn RJ, et al. Full Coverage for Preventive Medications
- 25. insurance systems. Journal of clinical epidemiology. Aug 2013;66(8 Suppl):S5-11. Choudhry NK, Shrank WH. Implementing randomized effectiveness trials in large
- 26 Devices (REMIND) trial. Contemporary clinical trials. Jul 2015;43:53-59. Randomized Evaluation to Measure Improvements in Non-adherence from Low-Cost Choudhry NK, Krumme AA, Ercole PM, et al. Rationale and design of the
- 27. myocardial infarction secondary preventive therapies. American heart journal. Jul FREEE trial: a randomized evaluation of first-dollar drug coverage for post-Choudhry NK, Brennan T, Toscano M, et al. Rationale and design of the Post-MI 2008;156(1):31-36.
- 28. 2009;157(4):613-619. based Generic Samples (SAMPLES) trial. American heart journal. Apr Shrank WH, Choudhry NK, Solomon DH, et al. Rationale and design of the Study Assessing the Effect of Cardiovascular Medications Provided as Low-cost, Evidence-
- 29. study. BMC endocrine disorders. 2012;12:20. and design of the multinational observational study assessing insulin use: the MOSAIc Polinski JM, Curtis BH, Seeger JD, Choudhry NK, Zagar A, Shrank WH. Rationale
- 30. reported measure of medication adherence. Medical care. Jan 1986;24(1):67-74. Morisky DE, Green LW, Levine DM. Concurrent and predictive validity of a self-
- 31. 2004;38(9):1363-1368. nonadherence with cardiovascular medications. The Annals of pharmacotherapy. Sep Shalansky SJ, Levy AR, Ignaszewski AP. Self-reported Morisky score for identifying
- 32. questionnaire (PHQ-2). Journal of psychosomatic research. Feb 2005;58(2):163-171 Lowe B, Kroenke K, Grafe K. Detecting and monitoring depression with a two-item
- 33 persistence in use of statin therapy in elderly patients. Jama. Jul 24-31 2002;288(4):455-461. Benner JS, Glynn RJ, Mogun H, Neumann PJ, Weinstein MC, Avorn J. Long-term
- 34. treatment intensification among patients with type 2 diabetes. Journal of general Patrick AR, Fischer MA, Choudhry NK, et al. Trends in insulin initiation and internal medicine. Feb 2014;29(2):320-327.
- 35 Modeling Techniques. Health services research. Apr 16 2015. Filling Predict Long-Term Adherence More Accurately Than High-Dimensional Franklin JM, Shrank WH, Lii J, et al. Observing versus Predicting: Initial Patterns of
- 36 approach to classifying and predicting long-term medication adherence. Medical care Sep 2013;51(9):789-796. Franklin JM, Shrank WH, Pakes J, et al. Group-based trajectory models: a new
- 37. of Statistics. 2001:1189-1232. Friedman JH. Greeding function approximation: a gradient boosting machine. Annals
- 38 2015;53(8):720-728. medication adherence thresholds and risk of hospitalization. Medical care. Aug Lo-Ciganic WH, Donohue JM, Thorpe JM, et al. Using machine learning to examine
- 39 Dec 2009;65(4):1254-1261. Czado C, Gneiting T, Held L. Predictive model assessment for count data. Biometrics



Clinical Study Protocol Appendix A

Drug Substance NA

Study Code D1843R00254

Edition Number

October 17, 2016 October 17, 2016

Protocol Dated

Signatures Appendix A

## ASTRAZENECA SIGNATURE(S)

### **Engagement in Diabetes Mellitus (ENGAGE-DM):** ENhancing outcomes through Goal Assessment and Generating

negotiated interviewing on disease control and medication adherence in patients with diabetes A 12-month study of the impact of combined shared-decision making and brief

This Clinical Study Protocol has been subjected to an internal AstraZeneca peer review

I agree to the terms of this study protocol/amendment.

site representative AstraZeneca Research and Developme

## ASTRAZENECA SIGNATURE(S)

### Engagement in Diabetes Mellitus (ENGAGE-DM): ENhancing outcomes through Goal Assessment and Generating

with diabetes negotiated interviewing on disease control and medication adherence in patients A 12-month study of the impact of combined shared-decision making and brief

This Clinical Study Protocol has been subjected to an internal AstraZeneca peer review

I agree to the terms of this study protocol/amendment

site representative AstraZeneca Research and Development

## ASTRAZENECA SIGNATURE(S)

### Engagement in Diabetes Mellitus (ENGAGE-DM): ENhancing outcomes through Goal Assessment and Generating

negotiated interviewing on disease control and medication adherence in patients with diabetes A 12-month study of the impact of combined shared-decision making and brief

This Clinical Study Protocol has been subjected to an internal AstraZeneca peer review.

I agree to the terms of this study protocol/amendment.

AstraZeneca Research and Development site representative

# SIGNATURE OF PRINCIPAL INVESTIGATOR

### **Engagement in Diabetes Mellitus (ENGAGE-DM): ENhancing outcomes through Goal Assessment and Generating**

with diabetes negotiated interviewing on disease control and medication adherence in patients A 12-month study of the impact of combined shared-decision making and brief

This Clinical Study Protocol has been subjected to an internal AstraZeneca peer review.

I agree to the terms of this amendment.

Signature: Centre No.: